CLINICAL TRIAL: NCT07386379
Title: The Effect of Propofol Infusion on Postoperative Nausea and Vomiting in Cardiac Surgery: A Prospective Observational Cohort Study
Brief Title: Propofol Infusion and PONV in Cardiac Surgery
Acronym: nausea vomitng
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yasemin Ozsahin, specialist, Istanbul University - Cerrahpasa
Other Study IDs: 1462022
Record Dates: First submitted 2025-12-08; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Nausea and Vomiting; Cardiovascular Surgical Procedures
Keywords: Postoperative Nausea and Vomiting; Propofol; Cardiac Surgical Procedures; Cardiovascular Surgical Procedures
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group H: High-Dose Propofol Group
- Group L: Low-Dose Propofol Group

SUMMARY:
The aim of this observational cohort study is to evaluate the effect of high-dose versus low-dose propofol infusion on the incidence of postoperative nausea and vomiting (PONV) in patients undergoing coronary artery bypass grafting (CABG). The study also seeks to assess the predictive performance of the Apfel and Koivuranta risk scores for PONV in the cardiac surgery population.

The primary objective of this study is to determine the impact of routinely administered high-dose propofol on the incidence and severity of PONV in CABG patients.

The secondary objective is to evaluate the need for antiemetic therapy during the intensive care unit stay.

The investigators will compare patients receiving high-dose propofol with those receiving low-dose propofol to determine whether the antiemetic effect of propofol is dose-dependent.

Participants will be asked to:

Allow PONV assessments to be performed during the first 24 hours postoperatively,

Provide permission for the collection of clinical data (including demographic characteristics, risk scores, opioid consumption, etc.) for research purposes.

DETAILED DESCRIPTION:
This research is designed as a prospective, observational cohort study to be conducted on patients undergoing open-heart surgery between November 2025 and March 2026. In the preoperative period, patients will be instructed to abstain from solid food intake after 24:00 on the night before surgery; consumption of non-alcoholic clear liquids will be allowed until two hours prior to the operation.

All procedures will be performed at the Istanbul University-Cerrahpaşa Cardiology Institute. Following the acquisition of written informed consent, all patients will be transferred to the operating room, where an 18G intravenous cannula will be inserted, and premedication will be administered with midazolam 0.03 mg/kg (IV).

Standard monitoring will include a five-lead electrocardiogram (ECG), heart rate assessment, invasive arterial blood pressure monitoring, and peripheral oxygen saturation measurement. All patients will undergo standard anesthesia induction with midazolam 0.15 mg/kg, fentanyl 10 µg/kg, and rocuronium 0.6 mg/kg (IV). Orotracheal intubation will be performed using an endotracheal tube of appropriate size according to the patient's age and sex.

Following intubation, mechanical ventilation will be initiated and adjusted to maintain an end-tidal carbon dioxide (EtCO₂) level between 35 and 45 mmHg. During anesthesia maintenance, the bispectral index (BIS) value will be kept within the 40-60 range. Total intravenous anesthesia (TIVA) will be maintained using propofol, fentanyl, and rocuronium infusions at the discretion of the attending anesthesiologist.

During surgery, all patients will be connected to a cardiopulmonary bypass (CPB) machine. After completion of graft placement and stabilization of vital signs, patients will be weaned from bypass. Postoperatively, patients will be transported to the intensive care unit (ICU) while still intubated, where mechanical ventilation will be continued and extubation will be performed according to their clinical condition.

Preoperative variables collected for the study will include age, sex, height, weight, body mass index (BMI), ASA physical status classification (ASA PS), smoking status, and history of postoperative nausea and vomiting (PONV) or motion sickness. Intraoperative variables will include type of surgical procedure, anesthesia technique, administered drug doses, PONV prophylaxis, duration of surgery, bypass time, and total anesthesia time.

In the postoperative period, duration of mechanical ventilation in the ICU will be recorded, and nausea/vomiting assessments will be conducted systematically by a blinded observer at 1, 2, 4, 8, and 24 hours after extubation.

Study Timeline Approximately 5-8 CABG procedures are performed weekly at the IUC Cardiology Institute operating suite. Taking into account patients who may be excluded, data collection from approximately 60 patients is expected to be completed within 3 months. An estimated additional 1-month period will be required for data analysis, interpretation, and manuscript preparation.

ELIGIBILITY:
Inclusion Criteria

Age ≥ 18 years

ASA physical status III

Elective coronary artery bypass grafting (CABG)

Surgery performed at Istanbul University-Cerrahpaşa, Cardiology Institute between November 2025 and March 2026

Exclusion Criteria

Gastrointestinal or central nervous system disorders within the past 3 months

Cochlear disorders associated with nausea and vomiting

Chronic opioid use

Advanced hepatic or renal disease

Alcohol or substance abuse

Left ventricular ejection fraction < 40%

Inability to be weaned from mechanical ventilation within 12 hours postoperatively

Postoperative morphine administration in the intensive care unit

Combined cardiac procedures (e.g., valve surgery)

Off-pump surgery

Emergency surgery

Reoperation due to bleeding or other complications

Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) classified as ASA III who are scheduled to undergo elective coronary artery bypass grafting (CABG) surgery at Istanbul University-Cerrahpaşa Cardiology Institute between November 2025 and March 2026. Patients with recent gastrointestinal or central nervous system disorders, cochlear conditions that may induce nausea or vomiting, chronic opioid use, severe hepatic or renal disease, alcohol or substance abuse, left ventricular ejection fraction <40%, prolonged postoperative mechanical ventilation (>12 hours), or postoperative morphine use in the ICU will be excluded. Additional exclusion criteria include combined cardiac procedures (e.g., valve surgery), off-pump CABG, emergency surgery, reoperation due to complications, and refusal to participate.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
the effect of high-dose propofol on PONV | 24 hours
  The primary objective of this study is to determine the impact of routinely administered high-dose propofol on the incidence and severity of PONV in CABG patients. Nausea and vomiting will be assessed at the 1st, 4th, 8th, and 24th postoperative hours. The severity will be classified as follows:
  None: No nausea or vomiting. Mild: Mild nausea or a single episode of vomiting, or nausea triggered by an external stimulus.
  Moderate: Two episodes of vomiting, nausea occurring without an external stimulus, and the need for one dose of antiemetic medication.
  Severe: Severe nausea, more than two episodes of vomiting, and the need for multiple doses of antiemetic medication.
  This follow-up and assessment method was adopted from the following study. Erkalp K, Kalekoglu Erkalp N, Sevdi MS, Korkut AY, Yeter H, Ege SS, Alagol A, Erden V. Gastric Decompression Decreases Postoperative Nausea and Vomiting in ENT Surgery. Int J Otolaryngol. 2014;2014:275860. doi: 10.1155/2014/275860.
the effect of high-dose propofol on PONV | 24 hours
  The primary objective of this study is to determine the impact of routinely administered high-dose propofol on the incidence and severity of PONV in CABG patients

SECONDARY OUTCOMES:
evaluate the need for antiemetic therapy in ICU | 24 hours
  The secondary objective is to evaluate the need for antiemetic therapy during the intensive care unit stay. Ondansetron requirement (in mg) will be recorded at the 1st, 4th, 8th, and 24th postoperative hours. Routine prophylactic antiemetic therapy will not be administered. Ondansetron will be administered only in patients classified as having moderate or severe nausea and vomiting according to the predefined severity scale, and the administered dose will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Ozsahin, Istanbul, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No